CLINICAL TRIAL: NCT00400777
Title: An Open-Label, Randomized, Multicenter Study to Evaluate the Efficacy of the Combination of Valsartan and Hydrochlorothiazide and Amlodipine in Hypertensive Patients Not Controlled With Valsartan and Hydrochlorothiazide
Brief Title: Efficacy and Safety of Valsartan, Hydrochlorothiazide and Amlodipine Combination Therapy in Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVEA489ABR01
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-06

CONDITIONS: Hypertension
Keywords: Valsartan; hydrochlorothiazide; amlodipine; hypertension; high blood pressure
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide; Amlodipine

INTERVENTIONS:
Drug: Valsartan, hydrochlorothiazide and amlodipine

SUMMARY:
This study is designed to evaluate the efficacy and safety of the combination valsartan with hydrochlorothiazide and amlodipine in hypertensive patients previously treated with valsartan with hydrochlorothiazide and remaining uncontrolled. A naturalistic approach will be taken comparing two different possible ways to achieve the higher dosage of the triple combination, i.e. 160 mg of valsartan and 25 mg of hydrochlorothiazide with amlodipine 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years of age
* Patients treated with up to two high blood pressure medications in a stable dose considered adequate by the investigator, for a minimum of two months, with blood pressure not controlled according to the following criteria:
* Systolic Blood Pressure ≥140 mmHg and/or Diastolic Blood Pressure ≥90 mmHg for low risk patients (no known target organ damage and without risk factor or presenting 1 - except Type 2 diabetes mellitus - risk factor);
* Systolic Blood Pressure ≥130 and/or Diastolic Blood Pressure ≥85 mmHg for medium risk patients (no known target organ damage and 2 or more risk factors - except Type 2 diabetes mellitus);
* Systolic Blood Pressure ≥130 and/or Diastolic Blood Pressure ≥80 mmHg for high risk patients (known target organ damage, and/or Type 2 diabetic patients and/or any clinically identifiable cardiovascular disease). OR
* Systolic Blood Pressure ≥160 mmHg and/or Diastolic Blood Pressure ≥100 mmHg at Visits 1 and 2 for previously untreated patients
* Patients previously treated but who stopped their medications will be considered untreated after one month without treatment
* Obs: -The target organ are: Brain, Heart, Kidney, Retina.
* The risk factors are: Smoking, Dyslipidemia, Age > 60 years old, and Family history of cardiovascular diseases (women < 65 years old and men < 55 years old

Exclusion Criteria:

* Systolic Blood Pressure ≥180 mmHg and/or Diastolic Blood Pressure ≥110 mmHg at Visit 1 or Visit 2
* Evidence of a secondary form of hypertension, to include coarctation of the aorta, primary hyperaldosteronism, renal artery stenosis, or pheochromocytoma
* Known Keith-Wagener grade III or IV hypertensive retinopathy
* History of hypertensive encephalopathy
* Cerebrovascular accident or myocardial infarction 12 months prior to Visit 1
* History of transient ischemic attack 12 months prior to Visit 1
* Percutaneous coronary intervention or coronary artery bypass graft surgery 12 months prior to Visit 1
* Diabetes mellitus type 1
* Diabetes mellitus type 2 under insulin treatment
* Poorly controlled type 2 diabetes mellitus
* History of heart failure Grade II - IV according to the NYHA classification
* Second or third degree heart block without a pacemaker
* Concomitant unstable angina pectoris
* Concomitant potentially life threatening arrhythmia or symptomatic arrhythmia
* Clinically significant valvular heart disease
* Women of child-bearing potential
* Pregnant or nursing (lactating) women
* Any surgical or medical condition which, at the discretion of the investigator, place the patient at higher risk from his/her participation in the study, or are likely to prevent the patient from complying with the requirements of the study or completing the trial period
* Additional protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2006-08; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reaching diastolic BP control, Proportion of patients reaching systolic BP control Percentage of diastolic responders,

SECONDARY OUTCOMES:
Mean change from study baseline in Diastolic Blood Pressure and in Systolic Blood Pressure after 4, 8 and 12 weeks of treatment
Mean change from study baseline in standing diastolic and systolic blood pressure after 4, 8 and 12 weeks of treatment
Safety and tolerability of the valsartan/HCTZ/amlodipine treatment algorithm strategy after 4, 8 and 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis AG, Study Chair — Sponsor GmbH
Locations (1):
- Novartis, Rio de Janeiro, Brazil